CLINICAL TRIAL: NCT04479423
Title: The Usage of Soda-Water in Gastric Preparation for Magnetically Controlled Capsule Endoscopy: A Prospective,Single Center,Randomized Controlled Study
Brief Title: The Usage of Soda-Water in Gastric Preparation for Magnetically Controlled Capsule Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Soda-water in MCE
Record Dates: First submitted 2020-07-06; First posted 2020-07-21 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Gastric Disease; Capsule Endoscopy
Keywords: capsule endoscopy; gastric distention; gastric transit time; clinical trial
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soda water (Experimental): 400ml soda water was drunk to obtain good vision before undergoing MCE examination.
  Interventions: Procedure: Soda-water instead of pure water to observe gastric filling
- water (No Intervention): 900ml clear water(100 ml water of simethicone solution was not included) was drunk to obtain good vision before undergoing MCE examination.

INTERVENTIONS:
Procedure: Soda-water instead of pure water to observe gastric filling — All patients underwent a bowel preparation that consisted of a low-residue diet for 24 hours, fluid intake, and ingestion of 2L polyethylene glycol-based electrolyte solution 12 hours before the examination. On the examination day, patients arrived at hospital in the morning after an over night fast (>8hours). Then they would be randomly assigned to controll group or soda group. 40 minutes before capsule ingestion, all patients swallowed 100ml clear water containing 50mg simethicone. During the period, patients were asked to have a proper walk to wash out bubbles. An additional 900ml pure water or 400ml soda-water was drunk to obtain good vision before undergoing MCE examination.
  Arms: Soda water

SUMMARY:
Magnetically controlled capsule endoscopy (MCE) is a noninvasive technique (90.4% sensitivity, 94.7% specificity and 93.4% accuracy) without requiring sedation or air insufflation, which makes it welcomed by most of participants. However, due to the large size of the stomach, clear views are obtained with the stomach distended. Participants were asked to drink 1000ml water for gastric preparation in a short time according to the standard procesure. It is hard for some participants especially the old and can cause discomfort. If the capsule stays in the stomach for a long time (>4 hours), it will affect the completion rate of small intestine examination and be inconvient to both of the endoscopist and patient.

It is a promising way to fill the stomach with carbonated drinks in some diagnosis and treatment methods. A study using carbonated drinks for gastric filling in the procedure of multi slice spiral computed tomography (MSCT) showed higher diagnostic rate for gastric cancer (85%VS80%). Rapid filling and absorption, greater comfort feeling and little pressure changes lead to higher acceptance of participants.

So, researchers have a novel idea using soda water to take place of pure water in the gastric preparation. The combination of gas and liquid in gastric filling greatly reduces the amount of fluid that participants need to drink, which makes the shorter preparation time and less feeling of fullness. In a pilot study before, investigators found the usage of soda water obtained similar gastric distention score and shorter gastric transit time (GTT) than standard preparation method.

This prospective, single blind, randomized controlleds trial aimed to prove the safety and efficiency of soda water in the process of gastric preparation and explore the impact on the follow-up small bowel examination.

DETAILED DESCRIPTION:
This is a prospective, single blind, randomized controlled clinical study approved by the Endoscopy Center of Changhai Hospital in Shanghai from July, 2020 to September,2020. Approval to carry out this study was granted by the Ethics Committee, Changhai Hospital, Naval Medical University.

According to the results of our pilot study, 252 participants(with 20% withdrawal rate) aged 18-75 will accept standard gastric preparation or gastric preparation with soda water randomly (ratio 1:1).All patient will provid written informed consent for this study before undergoing baseline MCE.

Investigators evaluated the feasibility of a novel gastric preparation methods regimens on gastric distention,gastric cleansing, feeling of fullness, diagnostic yield, satisfaction questionnaire, gastric transit time, small bowel transit time and completion rate. The safety were evaluated at two week after procedure for the occurance of adverse events. Investigators also plan to explore whether soda water can affect the subsequent examination of the small intestine, and the difficulty in intervention under special circumstances.

All participants underwent a bowel preparation that consisted of a low-residue diet for 24 hours, fluid intake, and ingestion of 2L polyethylene glycol-based electrolyte solution 12 hours before the examination. On the examination day, participants arrived at hospital in the morning after an over night fast (>8hours). Then they would be randomly assigned to controll group or soda group.

Control group:40 minutes before capsule ingestion, all participants swallowed 100ml clear water containing 50mg simethicone. During the period, participants were asked to have a proper walk to wash out bubbles. An additional 900ml clear water was drunk to obtain good vision before undergoing MCE examination.

Soda water group：Control group:40 minutes before capsule ingestion, all participants swallowed 100ml clear water containing 50mg simethicone. During the period, participants were asked to have a proper walk to wash out bubbles. An additional 400ml soda water was drunk to obtain good vision before undergoing MCE examination.

Then, the patient enter the examination room to finish the examination.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years and below 75 years of age
* Plan to undergo MCCG examination in Changhai Hospital

Exclusion Criteria:

* dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis, overt gastrointestinal bleeding, fistulas and strictures;
* history of gastrointestinal surgery or suspected delayed gastric emptying;
* Implanted metallic devices such aspacemakers, defibrillators, artificial heart valves or joint prostheses;
* Allergic to high molecular materials such as simethicone and streptozyme;
* Pregnancy or mentally ill person;
* currently participating in another clinical study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Gastric Filling of 0-5 minutes | 0-5 minutes after the capsule opened
  According to the extension of gastric plica on the great curvature, the score of gastric filling is ranged from 1 to 5 as excellent (smooth and basically no plica,score 5), good (the height of gastric plica <the distance between the adjacent gastric plica: score 4), fair (the height of gastric plica nearly same to the distance between the adjacent gastric plica: score 3),average (the height of gastric plica > the distance between the adjacent gastric plica: score 2) and poor (the folds gathered, and the gastric mucosa between plica is haedly to be seen, score 1).

SECONDARY OUTCOMES:
Fullness score | Before examination
  Fullness is the subjective feeling of patients assessed with visual analogue scale (VAS). VAS typically take the form of a straight line with two extreme states anchored at either end. In this study, it is a 100mm VAS with a question"How full do you feel?"anchored with "not at all full"at the left side and "as full as I have ever felt" at the right side. Patients will be asked to mark their feelings on the line. The distance (mm) between the far left and the marked point is the score of fullness. 0 represents no perception at all, 10 indicates pain and needs to be stopped immediately.
Satisfaction score of patients | After the procedure immediately
  All subjects were asked about tolerance of the procedure in the following areas using a questionnaire of Preprocedure Perception and Postprocedure Satisfaction, which including ease of swallowing, pain or discomfort experienced during and after the procedure, overall tolerability of the procedure, and overall convenience of the procedure (a score of 0-4,with 0 as the worst and 4 as the best respectively, ranged from 2 to 44).
Liquid for gastric refilling | During the procedure
  Count the numbers of patients who needs extra liguid which is used for better gastric distention during the examination procedure and how much they needed.
Gastric Examination Time (GET) | After the procedure(within 5 days)
  the time taken for the gastric examination to the endoscopist's satisfaction.
Gastric Cleanliness Score (GCS) | After the procedure(within 5 days)
  Six primary anatomical landmarks of the stomach (cardia, fundus, body, angulus, antrum, and pylorus) were recorded for evaluation. A 4-point grading scale was introduced to defne the cleanliness as excellent (no adherent mucus and foam: score 4), good (mild mucus and foam but do not obscure vision: score 3), fair (considerable amount of mucus or foam present precluding a completely reliable examination: score 2) and poor (large amount of mucus or foam residue needing water to clear it: score 1). GCS was the total scores of all six landmarks, ranging from 6 (completely unprepared) to 24 (perfect). GCS of≥18 was regarded as acceptable.
Transit Time | After the procedure(within 5 days)
  esophageal transit time (ETT),gastric transit time (GTT) and small bowel transit time (SBTT)
Diagnostic Yield (DY) | After the procedure(within 5 days)
  diagnostic yield including polyp, ulcer, gastric fundus varices, submucosal tumor, and carditis. The difuse lesions such as superfcial, atrophic, and erosive gastritis were defned as negative fndings.
Completion Rate (CR) | After the procedure(within 5 days)
  The completion of stomach was defined as the observation of cardia, fundus, body, angulus, antrum and pylorus and the completion of small bowel examination was defined as the ileocecal valve was photographed.The completion rate in each group was defined as the percentage of patients with a complete examination out of the total number of patients examined.
Gastric Filling score of 5-10 minutes | 5-10 minutes after the capsule opened
  According to the extension of gastric plica on the great curvature, the score of gastric filling is ranged from 1 to 5 as excellent (smooth and basically no plica,score 5), good (the height of gastric plica <the distance between the adjacent gastric plica: score 4), fair (the height of gastric plica nearly same to the distance between the adjacent gastric plica: score 3),average (the height of gastric plica > the distance between the adjacent gastric plica: score 2) and poor (the folds gathered, and the gastric mucosa between plica is haedly to be seen, score 1).

OTHER OUTCOMES:
Adverse events occurence rate | After 2-week follow-up period.
  The safety were evaluated at two week after procedure for any adverse events such as infection, pain, nausea, vomiting and capsule impaction or retention.

CONTACTS AND LOCATIONS:
Overall Officials: Liao Zhuan, MD, Study Chair — Department of Gastroenterology, Changhai Hospital, the Naval Medical University
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang YC, Pan J, Jiang X, Su XJ, Zhou W, Zou WB, Qian YY, Chen YZ, Liu X, Yu J, Yan XN, Zhao AJ, Li ZS, Liao Z. Repetitive Position Change Improves Gastric Cleanliness for Magnetically Controlled Capsule Gastroscopy. Dig Dis Sci. 2019 May;64(5):1297-1304. doi: 10.1007/s10620-018-5415-7. Epub 2018 Dec 17. PMID 30560329
- [Background] Stubbs RJ, Hughes DA, Johnstone AM, Rowley E, Reid C, Elia M, Stratton R, Delargy H, King N, Blundell JE. The use of visual analogue scales to assess motivation to eat in human subjects: a review of their reliability and validity with an evaluation of new hand-held computerized systems for temporal tracking of appetite ratings. Br J Nutr. 2000 Oct;84(4):405-15. doi: 10.1017/s0007114500001719. PMID 11103211
- [Background] Shimpo M, Akamatsu R. The effects of bowl size and portion size on food intake and fullness ratings in a sample of Japanese men. Public Health Nutr. 2018 Dec;21(17):3216-3222. doi: 10.1017/S1368980018001842. Epub 2018 Aug 6. PMID 30079861
- [Background] Jiang X, Qian YY, Liu X, Pan J, Zou WB, Zhou W, Luo YY, Chen YZ, Li ZS, Liao Z. Impact of magnetic steering on gastric transit time of a capsule endoscopy (with video). Gastrointest Endosc. 2018 Oct;88(4):746-754. doi: 10.1016/j.gie.2018.06.031. Epub 2018 Jul 11. PMID 30005825
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Liao Z, Duan XD, Xin L, Bo LM, Wang XH, Xiao GH, Hu LH, Zhuang SL, Li ZS. Feasibility and safety of magnetic-controlled capsule endoscopy system in examination of human stomach: a pilot study in healthy volunteers. J Interv Gastroenterol. 2012 Oct-Dec;2(4):155-160. doi: 10.4161/jig.23751. Epub 2012 Oct 1. PMID 23687601
- [Background] Westerhof J, Weersma RK, Koornstra JJ. Risk factors for incomplete small-bowel capsule endoscopy. Gastrointest Endosc. 2009 Jan;69(1):74-80. doi: 10.1016/j.gie.2008.04.034. Epub 2008 Aug 8. PMID 18691709
- [Background] Ohnhaus EE, Adler R. Methodological problems in the measurement of pain: a comparison between the verbal rating scale and the visual analogue scale. Pain. 1975 Dec;1(4):379-384. doi: 10.1016/0304-3959(75)90075-5. PMID 800639
- [Background] de Franchis R, Eisen GM, Laine L, Fernandez-Urien I, Herrerias JM, Brown RD, Fisher L, Vargas HE, Vargo J, Thompson J, Eliakim R. Esophageal capsule endoscopy for screening and surveillance of esophageal varices in patients with portal hypertension. Hepatology. 2008 May;47(5):1595-603. doi: 10.1002/hep.22227. PMID 18435461
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893